CLINICAL TRIAL: NCT04986904
Title: Optimizing Efficiency and Impact of Digital Health Interventions for Caregivers: A Mixed Methods Approach
Brief Title: Optimizing Efficiency and Impact of Digital Health Interventions for Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of Pittsburgh (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Kelly Shaffer, PhD, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR210255; R21TR003522 (NIH)
Record Dates: First submitted 2021-07-16; First posted 2021-08-03 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Family Caregivers; Insomnia; Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHUTi (Sleep Healthy Using the Internet) (Experimental): Participants will be assigned to the SHUTi (Sleep Healthy Using the Internet) online intervention. They will spend 1-2 hours each week for 6-9 weeks completing daily sleep diaries as well as interactive core content covering topics of sleep behaviors, sleep thoughts, sleep education, and relapse prevention. As users progress through the intervention, they will receive automated, tailored instructions for how to improve their sleep.
  Interventions: Behavioral: SHUTi (Sleep Healthy Using the Internet)

INTERVENTIONS:
Behavioral: SHUTi (Sleep Healthy Using the Internet) — Cognitive Behavioral Therapy for insomnia delivered online and metered out over 6 weeks in a fully automated, interactive, tailored web-based program
  Other Names: Cognitive-behavioral therapy for insomnia; CBT-I

SUMMARY:
The overall objective of this mixed-methods proposal is to answer the focused research question: What tailoring is necessary and sufficient to achieve optimal engagement with and efficacy of Sleep Healthy Using the Internet (SHUTi) for caregivers? The SHUTi program is a fully-automated Internet-delivered cognitive-behavioral therapy for insomnia (CBT-I) program. We will identify caregiving-related user- and environment characteristics that affect the use and impact of SHUTi, and other Internet interventions more broadly, for caregivers. We will recruit 100 high-intensity caregivers with insomnia to complete a baseline assessment of insomnia and caregiving context. Caregivers will then receive access to SHUTi in an open-label trial. At the end of the 9-week intervention period, caregivers will complete post-assessment and be categorized according to their level of engagement with the 6 SHUTi intervention lessons (or weekly "Cores"). We will test whether caregivers' engagement with SHUTi (i.e., being a non-user vs. incomplete user vs. complete user) is associated with their caregiving-related user characteristics (i.e., caregiving strain, self-efficacy, and guilt) and environment characteristics (i.e., proximity to care recipient; care recipient functional, cognitive, and behavioral status; caregiving tasks). Caregivers' barriers to and motivations for SHUTi engagement will be described from open-ended survey responses specific to participants' level of engagement as part of post-assessment. We will identify non-users' barriers to SHUTi adoption, the extent to which barriers were related to caregiving, and what modifications may have increased their motivation to try SHUTi. We will also identify users' (incomplete and complete) SHUTi usage barriers and motivations, the extent to which these were related to caregiving, and how tailoring may improve usage by increasing salience to caregivers. Thematic coding will also examine how caregivers' recommendations generalize to other evidence-based digital health interventions. Among caregivers using SHUTi, we will test whether the effects of SHUTi on cognitive mechanisms of change targeted by SHUTi (i.e., more adaptive sleep beliefs, internalized sleep locus of control) are associated with differences in caregiving-related user or environment characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Self-report providing high-intensity unpaid care (e.g., practical, medical, and/or emotional support) to a family member or "family-like" close individual, operationalized as a function of time spent caregiving and care task involvement.
* Self-report expecting to continue provide high-intensity care for at least another 3 months.
* Have access to any Internet-enabled device (computer, tablet, smartphone) and willing to be emailed about the study.
* Insomnia severity index score >= 10
* Residing in the United States or U.S. territory
* English literacy

Exclusion Criteria:

* Unusual average bed/wake times, including for shift work
* Current behavioral/psych treatment for insomnia
* Medical contraindication (Restless Leg Syndrome/Periodic Limb Movement Disorder, Obstructive Sleep Apnea, narcolepsy, parasomnia, dementia, Parkinson's, Huntington's, stroke, traumatic brain injury, brain infection/tumor, pregnancy/breastfeeding, hyperthyroidism, cancer, severe respiratory disease, epilepsy)
* Psychiatric contraindications (mania/hypomania, alcohol or substance abuse/dependence)
* Changes to prescription medications in the past 3 months (sleep, steroid, amphetamine, other wake-promoting)
* Severe computer literacy challenges

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
De-identified row-level data are available via data use agreement with the University of Virginia per institutional requirements; contact the primary investigator to initiate the contracting process.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
URL: https://bit.ly/SHUTiCARE-project

REFERENCES:
- [Background] Shaffer KM, Ritterband LM, You W, Buysse DJ, Mattos MK, Camacho F, Glazer JV, Klinger J, Donovan H. Single-Group Trial of an Internet-Delivered Insomnia Intervention Among Higher-Intensity Family Caregivers: Rationale and Protocol for a Mixed Methods Study. JMIR Res Protoc. 2022 Jan 12;11(1):e34792. doi: 10.2196/34792. PMID 35019846
- [Result] Shaffer KM, Ritterband LM, You W, Mattos MK, Buysse DJ, Glazer JV, Klinger J, Donovan H. Caregivers' Internet-Delivered Insomnia Intervention Engagement and Benefit: SHUTi-CARE Trial Primary Quantitative Analysis. Ann Behav Med. 2024 Oct 16;58(10):645-657. doi: 10.1093/abm/kaae031. PMID 38982942
- [Result] Shaffer KM, Perepezko K, Glazer JV, Mattos MK, Klinger J, Buysse DJ, Ritterband LM, Donovan H. Caregiver Experiences With an Internet-Delivered Insomnia Intervention: SHUTi-CARE Trial Primary Qualitative Analysis. Ann Behav Med. 2024 Oct 16;58(10):658-669. doi: 10.1093/abm/kaae041. PMID 38990523

RESULTS

PARTICIPANT FLOW:
Groups:
- SHUTi (Sleep Healthy Using the Internet): Participants were assigned to the SHUTi (Sleep Healthy Using the Internet) online intervention. They spent 1-2 hours each week for 6-9 weeks completing daily sleep diaries as well as interactive core content covering topics of sleep behaviors, sleep thoughts, sleep education, and relapse prevention. As users progressed through the intervention, they received automated, tailored instructions for how to improve their sleep.
  SHUTi (Sleep Healthy Using the Internet): Cognitive Behavioral Therapy for insomnia delivered online and metered out over 6 weeks in a fully automated, interactive, tailored web-based program
Period: Overall Study
Arm/Group | SHUTi (Sleep Healthy Using the Internet)
Started (This is the number of participants who were enrolled in the trial.) | 102
Completed Baseline Assessment (This is the number of participants who completed the baseline assessment, and were therefore provided access to the SHUTi intervention.) | 101 (One participant was lost-to-followup and did not complete the baseline assessment.)
Completed the 9-week Intervention Period (This is the number of participants who had access to SHUTi for the full 9-week intervention period, and were therefore counted towards the primary endpoint (i.e., level of engagement).) | 100 (One participant withdrew during the intervention period.)
Completed (This is the number of participants who completed post-assessment.) | 90 (Ten participants were lost-to-followup and did not complete post-assessment.)
Not Completed | 12
Not completed — Lost to Follow-up | 11
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Results are only reported from the 100 participants who received access to the SHUTi intervention for the full intervention period, and are therefore counted towards the primary endpoint (i.e., level of engagement). One participant who completed baseline but withdrew during the intervention period is excluded.
Arm/Group | SHUTi (Sleep Healthy Using the Internet)
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.82 (13.10)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 87
  Gender: Male | 11
  Gender: Other | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 94
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 14
  White | 79
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: SHUTi Engagement
Description: Level of SHUTi engagement: Core completion (i.e., nonuser [no cores completed], incomplete user [1-3 Cores], or complete user [4-6 Cores])
Time Frame: 9-week Post-assessment
Measure: Count of Participants; unit: Participants
Arm/Group | SHUTi (Sleep Healthy Using the Internet)
Number analyzed (Participants) | 100
Participants
  Non-User | 18
  Incomplete User | 22
  Complete User | 60

2. Secondary Outcome: Sleep-related Cognitions
Description: Dysfunctional Beliefs and Attitudes about Sleep; 16 items; sum scores range from 0 to 160 (higher scores indicate more dysfunctional attitudes and beliefs about sleep)
Time Frame: Baseline Pre-assessment and 9-week Post-assessment
Population: SHUTi Non-Users did not complete this measure at post-assessment. There were 6 SHUTi Incomplete Users who did not complete the post-assessment. All SHUTi Complete Users completed post-assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SHUTi Non-Users: Participants were assigned to the SHUTi (Sleep Healthy Using the Internet) online intervention. They spent 1-2 hours each week for 6-9 weeks completing daily sleep diaries as well as interactive core content covering topics of sleep behaviors, sleep thoughts, sleep education, and relapse prevention. As users progressed through the intervention, they received automated, tailored instructions for how to improve their sleep.
  SHUTi (Sleep Healthy Using the Internet): Cognitive Behavioral Therapy for insomnia delivered online and metered out over 6 weeks in a fully automated, interactive, tailored web-based program.
  Participants were classified as non-users if they did not complete any of the six SHUTi Cores.
- SHUTi Incomplete Users: Participants were assigned to the SHUTi (Sleep Healthy Using the Internet) online intervention. They spent 1-2 hours each week for 6-9 weeks completing daily sleep diaries as well as interactive core content covering topics of sleep behaviors, sleep thoughts, sleep education, and relapse prevention. As users progressed through the intervention, they received automated, tailored instructions for how to improve their sleep.
  SHUTi (Sleep Healthy Using the Internet): Cognitive Behavioral Therapy for insomnia delivered online and metered out over 6 weeks in a fully automated, interactive, tailored web-based program.
  Participants were classified as users if they completed one to three of the six SHUTi Cores.
- SHUTi Complete Users: Participants were assigned to the SHUTi (Sleep Healthy Using the Internet) online intervention. They spent 1-2 hours each week for 6-9 weeks completing daily sleep diaries as well as interactive core content covering topics of sleep behaviors, sleep thoughts, sleep education, and relapse prevention. As users progressed through the intervention, they received automated, tailored instructions for how to improve their sleep.
  SHUTi (Sleep Healthy Using the Internet): Cognitive Behavioral Therapy for insomnia delivered online and metered out over 6 weeks in a fully automated, interactive, tailored web-based program.
  Participants were classified as users if they completed four or more of the six SHUTi Cores.
Arm/Group | SHUTi Non-Users | SHUTi Incomplete Users | SHUTi Complete Users
Number analyzed (Participants) | 18 | 22 | 60
score on a scale
  Baseline | 92.61 (31.54) | 92.68 (18.20) | 86.08 (27.04)
  Post-Assessment: number analyzed (Participants) | 0 | 16 | 60
  Post-Assessment |  | 61.12 (36.20) | 54.82 (30.08)

3. Secondary Outcome: Sleep Self-efficacy
Description: Sleep Locus of Control Scale with two subscales:
  1. a 5-item subscale for internal locus of control; summed scores per scale range from 5 to 30 (higher scores indicate higher belief in the locus of control measured; higher internal sleep locus of control is a better outcome)
  2. a 3-item subscale for external locus of control; summed scores per scale range from 3 to 18 (higher scores indicate higher belief in the locus of control measured; lower external sleep locus of control is a better outcome)
Time Frame: Baseline Pre-assessment and 9-week Post-assessment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHUTi Non-Users | SHUTi Incomplete Users | SHUTi Complete Users
Number analyzed (Participants) | 18 | 22 | 60
score on a scale
  Baseline Sleep Locus of Control - Internal | 17.06 (4.49) | 14.77 (4.06) | 15.02 (4.85)
  Post-Assessment Sleep Locus of Control - Internal: number analyzed (Participants) | 0 | 16 | 60
  Post-Assessment Sleep Locus of Control - Internal |  | 15.94 (6.39) | 16.93 (5.12)
  Baseline Sleep Locus of Control - External | 9.11 (4.14) | 8.14 (3.17) | 8.68 (3.72)
  Post-Assessment Sleep Locus of Control - External: number analyzed (Participants) | 0 | 16 | 60
  Post-Assessment Sleep Locus of Control - External |  | 6.69 (3.09) | 6.75 (3.00)

4. Other Pre Specified Outcome: Open-ended Feedback on SHUTi
Description: Non-users' post-assessment will include an open-ended survey regarding barriers to SHUTi adoption, the extent to which barriers were related to caregiving, and what modifications may have increased their motivation to try SHUTi. Users' (i.e., incomplete and complete) post-assessment will include an open-ended survey assessing SHUTi usage barriers and motivations, the extent to which these were related to caregiving, and how tailoring may improve usage by increasing salience to caregivers.
Time Frame: 9-week Post-assessment
Reporting Status: Not Posted

5. Other Pre Specified Outcome: SHUTi Evaluation
Description: Items from the Internet Intervention Utility, Evaluation, and Adherence questionnaire assess users' perceived usability, acceptability, and perceived efficacy of SHUTi as well as barriers to program use
Time Frame: 9-week Post-assessment
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Caregiving Strain
Description: Pearlin Stress Scale - Overload subscale; 4 items; averaged scores range from 1 to 4 (higher scores indicate greater perceived burden)
Time Frame: Baseline Pre-assessment and 9-week Post-assessment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Insomnia Symptom Severity
Description: Insomnia severity index; 2 items; summed scores range from 0 to 8 (higher scores indicate more severe insomnia symptoms)
Time Frame: Baseline Pre-assessment and 9-week Post-assessment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Sleep Onset Latency (SOL)
Description: Data collected from sleep diary: Time fell asleep - Time attempting to fall asleep
Time Frame: Baseline Pre-assessment and 9-week Post-assessment
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Wake After Sleep Onset (WASO)
Description: Data collected from sleep diary: Total time awake between time feel asleep and final morning waking
Time Frame: Baseline Pre-assessment and 9-week Post-assessment
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Perceived Sleep Quality
Description: Data collected from sleep diary: Nightly rating of perceived sleep quality from very poor to very good
Time Frame: Baseline Pre-assessment and 9-week Post-assessment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | SHUTi (Sleep Healthy Using the Internet)
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT04986904/Prot_SAP_002.pdf
  • Informed Consent Form (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT04986904/ICF_001.pdf